CLINICAL TRIAL: NCT02804204
Title: Analysis of Circulant Rheumatoid Factor, Cyclic Citrullinated Anti-peptide Anti-bodies and Albumin as a Potential Predictor in the Response to the Treatment With Anti-TNF in Patients With Rheumatoid Arthritis
Brief Title: Serum Biomarkers Analysis in Patients With AR Treated With Anti-TMF
Acronym: AROMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: SMB-CZP- 2014-03
Record Dates: First submitted 2016-06-08; First posted 2016-06-17 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2016-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anti-TNF
  Interventions: Drug: Anti-TNF

INTERVENTIONS:
Drug: Anti-TNF

SUMMARY:
Multicenter, prospective, observational study for evaluating if circulant rheumatoid factor, cyclic citrullinated anti-peptide anti-bodies and albumin can be used as potential predictors in the response to the treatment with anti-TNF in patients with rheumatoid arthritis after 24 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Over 18 years old
* Diagnosis of rheumatoid arthritis according to ACR criteria
* Patients that initiate treatment with anti-TNF drugs according to clinical practice, both in naïve anti-TNF patients and patients after first anti-TNF failure
* Patients able to follow the protocol requirements
* Patients that signed the informed consent

Exclusion Criteria:

* Patients with known hypersensitivity to investigational products
* Patients with tuberculosis, or severe infections like sepsis or opportunistic infections
* Patients with moderate/severe cardiac insufficiency (NHYA classification Class III/IV)
* Patients that according to the investigator criteria can not participate in the study or complete the study questionnaires
* Pregnant or fertile woman that does not use a contraception method

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis according to the ACR criteria
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Anti-TNF treatment response based on circulant rheumatoid factor | 24 weeks
Anti-TNF treatment response based on circulant cyclic citrullinated anti-peptide antibodies. | 24 weeks

CONTACTS AND LOCATIONS:
Locations (19):
- Spain (19):
  - Hospital San Cecilio, Granada, Andalusia
  - Hospital Carlos Haya, Málaga, Andalusia
  - Hospital Virgen del Rocio, Seville, Andalusia
  - Hospital Son LLatzer, Palma de Mallorca, Balearic Islands
  - Hospital de Basurto, Bilbao, Basque Country
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Canary Islands
  - Hospital Marques de Valdecilla, Santander, Cantabria
  - Hospital de Guadalajara, Guadalajara, Castille-La Mancha
  - Hospital Vall d'Hebron, Barcelona, Catalonia
  - Clínic de Barcelona, Barcelona, Catalonia
  - Hospital de Santa Creu i Sant Pau, Barcelona, Catalonia
  - Hospital de Bellvitge, L'Hospitalet de Llobregat, Catalonia
  - Hospital Moises Broggi, Sant Joan Despí, Catalonia
  - Complexo Hospitalaria A Coruña, A Coruña, Galicia
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital Infanta Sofía, Madrid, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital Puerta de Hierro, Madrid, Madrid
  - Hospital Virgen de la Arreixaca, Murcia, Murcia